CLINICAL TRIAL: NCT01835470
Title: A Phase III, Multicenter, Open-Label Study to Assess Efficacy, Safety, Pharmacokinetics and Immunogenicity of Abatacept Administered Intravenously in Japanese Children and Adolescents With Active Juvenile Idiopathic Arthritis Who Have a History of an Inadequate Response or Intolerance to Methotrexate or Biologics
Brief Title: Efficacy, Safety, Pharmacokinetics and Immunogenicity Study of Abatacept Administered Intravenously to Treat Active Polyarticular-course Juvenile Idiopathic Arthritis in Japan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM101-365
Record Dates: First submitted 2013-04-17; First posted 2013-04-19 (Estimated); Results first posted 2017-01-11 (Estimated); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abatacept (Experimental): Abatacept 10 mg/kg (for body weight less than 75 kg), 750 mg (for body weight between 75 and 100 kg), and 1g (for body weight above 100kg) intravenous infusion on Week 0 (Day 1), Week 2 (Day 15), Week 4 (Day 29) and every 4 weeks (28 days) thereafter up to the end of the study
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept
  Other Names: BMS-188667; ONO-4164

SUMMARY:
The purpose of this study is to assess the efficacy of Abatacept after intravenous administration in Japanese children and adolescents with active juvenile idiopathic arthritis who have a history of an inadequate response or intolerance to Methotrexate or biologics

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have a history of an inadequate therapeutic response or intolerance in the opinion of the examining physician to at least one biologics or Methotrexate (MTX).
* Diagnosis of Juvenile Idiopathic Arthritis (JIA) by International League of Associations for Rheumatology (ILAR) criteria as oligoarticular, polyarticular Rheumatoid Factor (RF+), polyarticular (RF-), or systemic with a polyarticular-course.
* Men and women, ages 4 to 17 years, inclusive at enrollment.
* Subjects must have a history of at least 5 joints with active disease and must have currently active articular disease as defined by:

  1. ≥2 active joints (e.g. presence of swelling, or if no swelling is present, limitation of motion (LOM) accompanied by pain, tenderness, or both) at screening and at Week 0 (Day 1).
  2. ≥2 joints with LOM at screening and at Week 0 (Day 1).

Exclusion Criteria:

* Systemic onset JIA with any of the following manifestations within the last 6 months prior to enrollment: intermittent fever due to JIA, rheumatoid rash, hepatosplenomegaly, pleuritis, pericarditis, or macrophage activation syndrome.
* Presence of any other rheumatic disease or major chronic infectious/inflammatory/immunologic disease (e.g. inflammatory bowel disease, psoriatic arthritis, spondyloarthropathy, hypogammaglobulinemia, or systemic lupus erythematosus, etc.)

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2013-08-09 (Actual); Primary Completion 2015-11-24 (Actual); Study Completion 2018-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (11):
- Japan (11):
  - Local Institution, Oobu-shi, Aichi-ken
  - Local Institution, Sapporo, Hokkaido
  - Local Institution, Kobe, Hyōgo
  - Local Institution, Kagoshima, Kagoshima-ken
  - Local Institution, Yokohama, Kanagawa
  - Local Institution, Sendai, Miyagi
  - Local Institution, Niigata, Niigata
  - Local Institution, Nakagami-gun, Okinawa
  - Local Institution, Takatsuki-shi, Osaka
  - Local Institution, Bunkyo-ku, Tokyo
  - Local Institution, Shinjuku-ku, Tokyo

REFERENCES:
- [Derived] Hara R, Umebayashi H, Takei S, Okamoto N, Iwata N, Yamasaki Y, Nakagishi Y, Kizawa T, Kobayashi I, Imagawa T, Kinjo N, Amano N, Takahashi Y, Mori M, Itoh Y, Yokota S. Intravenous abatacept in Japanese patients with polyarticular-course juvenile idiopathic arthritis: results from a phase III open-label study. Pediatr Rheumatol Online J. 2019 Apr 30;17(1):17. doi: 10.1186/s12969-019-0319-4. PMID 31039807
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 23 participants were enrolled and 20 participants were treated. Reason for non-treatment was that 3 participants no longer met study criteria.
Period: Short Term Treatment Period (to Week 16)
Arm/Group | Abatacept
Started | 20
Completed | 20
Not Completed | 0
Period: Long Term Treatment Period
Arm/Group | Abatacept
Started | 20
Completed | 16 (Completed LT period)
Not Completed | 4
Not completed — Subject Request to Discontinue | 1
Not completed — Lack of Efficacy | 3

BASELINE CHARACTERISTICS:
Population: All Treated Participants: All participants who received at least one dose of study medication
Arm/Group | Abatacept
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.2 (3.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 20
Region of Enrollment [Number; unit: Participants]
  Japan | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing a American College of Rheumatology (ACR) Pediatric 30 Response at Week 16
Description: American College of Rheumatology (ACR) pediatric (PED) 30 response was defined as '≥30% improvement' and '≥3 of the 6 Juvenile Idiopathic Arthritis (JIA) core set' and ≥30% worsening in not more than 1 of the 6 JIA core set variables. JIA core set variables defined as the number of active joints, number of joints with Limit of Motion (LOM), physician's global assessment of disease severity, patient global assessment of overall well being, parent assessment of physical function, and acute phase reactant value. A non-responder imputation was applied.
Time Frame: Week 16 (Day 113)
Population: All Treated Participants: All participants who received at least one dose of study medication
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Abatacept
Number analyzed (Participants) | 20
percentage of participants | 90.0 [68.3 to 98.8]

2. Secondary Outcome: Percentage of Participants Experiencing a American College of Rheumatology Pediatric 50, 70, 90 Response or Inactive Disease at Week 16
Description: ACR PED 50 response is defined as '≥50% improvement' and '≥3 of the 6 Juvenile Idiopathic Arthritis (JIA) core set' and ≥30% worsening in not more than 1 of the 6 JIA core set variables. ACR PED 70 response is defined as '≥70% improvement' and '≥3 of the 6 JIA core set' and ≥30% worsening in not more than 1 of the 6 JIA core set variables. ACR PED 90 response is defined as '≥90% improvement' and '≥3 of the 6 JIA core set' and ≥30% worsening in not more than 1 of the 6 JIA core set variables. Inactive disease status is defined as no active joints, physician's global assessment of disease severity equal or less than 10mm and C-reactive protein (CRP) within normal limits (0.3 mg/dL). A non-responder imputation is applied. mm=millimeter; mg/dL=milligrams/deciliter
Time Frame: Week 16 (Day 113)
Population: All Treated Participants: All participants who received at least one dose of study medication
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Abatacept
Number analyzed (Participants) | 20
percentage of participants
  ACR PED 50 | 75.0 [50.9 to 91.3]
  ACR PED 70 | 70.0 [45.7 to 88.1]
  ACR PED 90 | 35.0 [15.4 to 59.2]
  Inactive Disease | 25.0 [8.7 to 49.1]

3. Secondary Outcome: Median Percentage of Improvement From Baseline in Physical Function as Assessed by the Childhood Health Assessment Questionnaire (CHAQ) Disability Index at Week 16
Description: Physical function was evaluated using the disability section of the Childhood Health Assessment Questionnaire (CHAQ). The questionnaire was derived from the adult HAQ. The disability section assessed physical functions in 8 domains: dressing and grooming, arising, eating, walking, hygiene, reach, grip and common activities. The questions were evaluated on a 4-point scale: 0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty and 3 =unable to do. Higher scores indicate greater dysfunction. A disability index was calculated as the mean of the 8 functional scales. The percentage of Improvement from baseline was calculated using the following equation: (Baseline value - Post-baseline value) / Baseline value x 100.
Time Frame: Week 16 (Day 113)
Population: All Treated Participants: All participants who received at least one dose of study medication
Measure: Median (Inter-Quartile Range); unit: percentage of improvement from baseline
Arm/Group | Abatacept
Number analyzed (Participants) | 20
percentage of improvement from baseline | 43.18 [0.00 to 100.00]

4. Secondary Outcome: Number of Participants With Death, Serious Adverse Events (SAEs), Drug-Related SAEs, Discontinuation Due to Drug-Related SAEs, Drug-Related Adverse Events (AEs), and Discontinuation Due to Drug-Related AEs During the Short Term Period
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. SAEs also include hospitalizations for elective surgical procedures. Drug-related=related or missing relationship to study drug. Data includes all events from the date of the first dose of the study drug up to 56 days post the last dose of the study drug in the short-term period or start of the long-term period, whichever occurred first.
Time Frame: Day 1 up to 56 days post Week 16 (Day 113); approximately 6 months
Population: All Treated Participants: All participants who received at least one dose of study medication
Measure: Number; unit: participants
Arm/Group | Abatacept
Number analyzed (Participants) | 20
participants
  Death | 0
  SAEs | 2
  Drug-Related SAEs | 1
  Discontinuation Due to Drug-Related SAEs | 0
  Drug-Related AEs | 5
  Discontinuation Due to Drug-Related AEs | 0

5. Secondary Outcome: Maximum Observed Concentration (Cmax) of Abatacept During the Short Term Period
Description: Cmax was obtained from the serum concentration versus time data after intravenous administration of abatacept. Blood samples were collected at 0 hour (pre-dose) on Days 15 and 29 and at 0 hour (pre-dose) and 0.5 hours (post dose) on Days 57, 85, and 113. A blood sample was also collected on an interim visit that occurred on any day between Day 92 and Day 110. ug/mL=micrograms/milliliter
Time Frame: 9 time points up to Week 16 (Day 113)
Population: Pharmacokinetic (PK) Analysis Population: All participants who received at least one dose of study medication and who had at least one adequate PK result reported after start of study medication. The 'n' signifies those participants who received study drug and were evaluated for this measure (each group respectively).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Abatacept
Number analyzed (Participants) | 20
ug/mL
  Day 57 | 163.13 (26.22)
  Day 85 | 172.43 (23.15)
  Day 113 | 167.85 (18.42)

6. Secondary Outcome: Trough Observed Concentration (Ctrough) of Abatacept During the Short Term Period
Description: Blood samples were collected at 0 hour (pre-dose) on Days 15 and 29 and at 0 hour (pre-dose) and 0.5 hours (post dose) on Days 57, 85, and 113. A blood sample was also collected on an interim visit that occurred on any day between Day 92 and Day 110. ug/mL=micrograms/milliliter
Time Frame: 9 time points up to Week 16 (Day 113)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Abatacept
Number analyzed (Participants) | 20
ug/mL
  Day 15: number analyzed (Participants) | 18
  Day 15 | 25.50 (27.61)
  Day 29: number analyzed (Participants) | 17
  Day 29 | 38.64 (29.08)
  Day 57 | 17.24 (36.63)
  Day 85: number analyzed (Participants) | 18
  Day 85 | 16.79 (40.01)
  Day 113: number analyzed (Participants) | 19
  Day 113 | 15.56 (36.61)

7. Secondary Outcome: Number of Participants With Positive Immunogenicity During the Short Term Period
Description: A positive immunogenicity response for 'Cytotoxic T-lymphocyte antigen (CTLA4), Immunoglobulin (Ig)', 'Ig and/or Junction Region', respectively = (1) missing baseline immunogenicity measurement and positive analytical laboratory reported immunogenicity response post-baseline (2) negative baseline immunogenicity response and positive analytical laboratory reported immunogenicity response post-baseline (3) positive baseline immunogenicity response and positive analytical laboratory reported immunogenicity response post-baseline with titer value strictly greater than the baseline titer value. Assessment based on assay cutpoint value. Serum samples were collected prior to study medication at Week 0 (Day 1), Week 8 (Day 57), and Week 16 (Day 113) in the short term period. Participants who early discontinued from the study or complete and did not switch to commercial abatacept had a serum sample collected on final visit or early termination visit, 28, 84 and 168 days after the last dose.
Time Frame: Day 1 up to Week 16 (Day 113)
Population: Immunogenicity analysis population: All participants who received at least one dose of study medication and who had at least one immunogenicity result reported after start of study medication
Measure: Number; unit: participants
Arm/Group | Abatacept
Number analyzed (Participants) | 20
participants | 0

ADVERSE EVENTS:
Time Frame: During the cumulative period which is from the first dose date up to 56 days beyond the last dose of study medication in the LT period for participants entering the LT or up to 56 days beyond the last dose of study medication in the ST period for participants not entering the LT period
Description: From September 2013 to July 2018 (approximately 61 months)
Arm/Group | IV ABATACEPT
Serious Adverse Events (participants affected / at risk) | 6/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IV ABATACEPT (N=20)
ENTEROCOLITIS VIRAL (Infections and infestations) | 1
GASTROENTERITIS (Infections and infestations) | 1
VARICELLA (Infections and infestations) | 1
VIRAL TONSILLITIS (Infections and infestations) | 1
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1
JUVENILE IDIOPATHIC ARTHRITIS (Musculoskeletal and connective tissue disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IV ABATACEPT (N=20)
DRY EYE (Eye disorders) | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2
APHTHOUS ULCER (Gastrointestinal disorders) | 2
CONSTIPATION (Gastrointestinal disorders) | 2
DIARRHOEA (Gastrointestinal disorders) | 5
NAUSEA (Gastrointestinal disorders) | 4
STOMATITIS (Gastrointestinal disorders) | 7
TOOTHACHE (Gastrointestinal disorders) | 2
VOMITING (Gastrointestinal disorders) | 3
PYREXIA (General disorders) | 4
SEASONAL ALLERGY (Immune system disorders) | 5
ANGULAR CHEILITIS (Infections and infestations) | 2
BRONCHITIS (Infections and infestations) | 5
CONJUNCTIVITIS (Infections and infestations) | 3
ENTEROCOLITIS VIRAL (Infections and infestations) | 2
GASTROENTERITIS (Infections and infestations) | 4
INFLUENZA (Infections and infestations) | 10
NASOPHARYNGITIS (Infections and infestations) | 17
PHARYNGITIS (Infections and infestations) | 12
RHINITIS (Infections and infestations) | 3
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4
VIRAL PHARYNGITIS (Infections and infestations) | 3
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 2
CONTUSION (Injury, poisoning and procedural complications) | 6
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 7
SKIN ABRASION (Injury, poisoning and procedural complications) | 2
INFLUENZA B VIRUS TEST POSITIVE (Investigations) | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2
MYALGIA (Musculoskeletal and connective tissue disorders) | 2
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2
TENDONITIS (Musculoskeletal and connective tissue disorders) | 2
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
HEADACHE (Nervous system disorders) | 7
COUGH (Respiratory, thoracic and mediastinal disorders) | 3
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 3
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 2
UPPER RESPIRATORY TRACT INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 6
ACNE (Skin and subcutaneous tissue disorders) | 5
ALOPECIA (Skin and subcutaneous tissue disorders) | 2
DERMATITIS (Skin and subcutaneous tissue disorders) | 2
DRY SKIN (Skin and subcutaneous tissue disorders) | 2
ECZEMA (Skin and subcutaneous tissue disorders) | 2
PURPURA (Skin and subcutaneous tissue disorders) | 2
RASH (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.